CLINICAL TRIAL: NCT04164082
Title: Phase II Trial of Intravesical Gemcitabine and MK-3475 (Pembrolizumab) in the Treatment of Patients With BCG-Unresponsive Non-Muscle Invasive Bladder Cancer
Brief Title: Testing the Addition of an Anti-cancer Drug, Pembrolizumab, to the Usual Intravesical Chemotherapy Treatment (Gemcitabine) for the Treatment of BCG-Unresponsive Non-muscle Invasive Bladder Cancer
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2019-07573; NCI-2019-07573 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); A031803 (Other: Alliance for Clinical Trials in Oncology); A031803 (Other: CTEP); U10CA180821 (NIH)
Record Dates: First submitted 2019-11-14; First posted 2019-11-15 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Bladder Flat Urothelial Carcinoma In Situ; Non-Muscle Invasive Bladder Urothelial Carcinoma; Stage 0a Bladder Cancer AJCC v8; Stage 0is Bladder Cancer AJCC v8; Stage I Bladder Cancer AJCC v8
MeSH Terms: conditions — Urinary Bladder Neoplasms | interventions — Biopsy; Specimen Handling; Cystoscopy; Gemcitabine; Magnetic Resonance Spectroscopy; pembrolizumab; Transurethral Resection of Bladder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (pembrolizumab, gemcitabine hydrochloride) (Experimental): INDUCTION: Patients receive pembrolizumab IV over 25-40 minutes on day 1 of cycles 1-4. Patients also receive gemcitabine hydrochloride intravesically on days 1, 8 and 15 of cycles 1 and 2. Treatment repeats every 3 weeks for 4 cycles in the absence of disease progression or unacceptable toxicity.
  MAINTENANCE: Beginning cycle 5, patients with no evidence of disease after induction receive pembrolizumab IV over 25-40 minutes and gemcitabine intravesically on day 1 of each cycle. Treatment repeats every 3 weeks for 12 cycles in the absence of disease progression or unacceptable toxicity.
  Additionally, patients with T1 tumors undergo a re-staging TURBT within 60 days of registration. Patients also undergo urine and blood sample collection, bladder biopsy, cystoscopy, CT and MRI throughout the study.
  Interventions: Procedure: Biopsy Procedure; Procedure: Biospecimen Collection; Procedure: Computed Tomography; Procedure: Cystoscopy; Drug: Gemcitabine Hydrochloride; Procedure: Magnetic Resonance Imaging; Biological: Pembrolizumab; Procedure: Transurethral Resection of Bladder Tumor

INTERVENTIONS:
Procedure: Biopsy Procedure — Undergo bladder biopsy
  Other Names: Biopsy; BIOPSY_TYPE; Bx
Procedure: Biospecimen Collection — Undergo urine and blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Computed Tomography — Undergo CT
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; Diagnostic CAT Scan; Diagnostic CAT Scan Service Type; tomography
Procedure: Cystoscopy — Undergo cystoscopy
  Other Names: CS
Drug: Gemcitabine Hydrochloride — Given intravesically
  Other Names: dFdCyd; Difluorodeoxycytidine Hydrochloride; Gemcitabine HCI; Gemzar; LY 188011; LY-188011; LY188011
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance; Magnetic Resonance Imaging (MRI); Magnetic resonance imaging (procedure); Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; MRIs; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging; sMRI; Structural MRI
Biological: Pembrolizumab — Given IV
  Other Names: BCD-201; GME 751; GME751; Keytruda; Lambrolizumab; MK 3475; MK-3475; MK3475; Pembrolizumab Biosimilar BCD-201; Pembrolizumab Biosimilar GME751; Pembrolizumab Biosimilar QL2107; Pembrolizumab Biosimilar RPH-075; Pembrolizumab Biosimilar SB27; QL2107; RPH 075; RPH-075; RPH075; SB 27; SB-27; SB27; SCH 900475; SCH-900475; SCH900475
Procedure: Transurethral Resection of Bladder Tumor — Undergo TURBT
  Other Names: Transurethral resection (TURBT); TURBT

SUMMARY:
This phase II trial studies the effect of adding pembrolizumab to gemcitabine in treating patients with non-muscle invasive bladder cancer whose cancer does not respond to Bacillus Calmette-Guerin (BCG) treatment. Chemotherapy drugs, such as gemcitabine, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Immunotherapy with monoclonal antibodies, such as pembrolizumab, may help the patient's immune system attack the cancer, and may interfere with the ability of tumor cells to grow and spread. Adding pembrolizumab to gemcitabine may delay the return of BCG-unresponsive bladder cancer for longer period compared to gemcitabine alone.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Estimate the 6-month complete response rate of treatment with intravesical gemcitabine hydrochloride (gemcitabine) in combination with MK-3475 (pembrolizumab) in patients with Bacillus Calmette-Guerin (BCG)-unresponsive non-muscle invasive bladder cancer (NMIBC) that have a carcinoma in situ (CIS) component.

II. Estimate the 18 month event-free survival (EFS) rate for all patients with BCG-unresponsive NMIBC receiving intravesical gemcitabine in combination with MK-3475 (pembrolizumab).

SECONDARY OBJECTIVES:

I. To characterize the safety profile of the combination of intravesical gemcitabine with MK-3475 (pembrolizumab) with BCG-unresponsive NMIBC (CIS or high grade Ta and T1 with or without a CIS component).

II. To estimate progression-free survival (PFS) of patients with BCG-unresponsive NMIBC treated with intravesical gemcitabine in combination with MK-3475 (pembrolizumab).

III. To estimate overall survival (OS) of patients with BCG-unresponsive NMIBC treated with intravesical gemcitabine in combination with MK-3475 (pembrolizumab).

IV. To estimate cystectomy-free survival of patients with BCG-unresponsive NMIBC treated with intravesical gemcitabine in combination with MK-3475 (pembrolizumab).

V. To estimate recurrence-free survival (RFS) for patients with a CIS component only and those without a CIS component.

EXPLORATORY OBJECTIVES:

I. To assess correlation between tumor mutation burden (TMB) and EFS and 6-month complete response (CR) rate.

II. To assess correlation between specific genomic alterations (single nucleotide variant [SNV] and copy number gains/loss) and EFS and 6-month complete response rate.

III. To assess correlation between APOBEC mutational signature and EFS and 6-month complete response rate.

IV. To assess correlation between immune gene signatures (IGS) and EFS and 6-month complete response rate.

V. To assess correlation between PD-L1 ribonucleic acid (RNA) levels and EFS and 6-month complete response rate.

VI. To assess correlation between RNA molecular subtype and EFS and 6-month complete response rate.

VII. To assess correlation between intratumoral T-cell receptor (TCR) clonality and EFS and 6-month complete response rate.

VIII. To assess correlation between changes in peripheral blood TCR clonality and EFS and 6-month complete response rate.

IX. To assess EFS in patients with urine cell free deoxyribonucleic acid (DNA) (cfDNA) + versus (vs.) patients with cfDNA.

OUTLINE:

INDUCTION: Patients receive pembrolizumab intravenously (IV) over 25-40 minutes on day 1 of cycles 1-4. Patients also receive gemcitabine hydrochloride intravesically on days 1, 8 and 15 of cycles 1 and 2. Treatment repeats every 3 weeks for 4 cycles in the absence of disease progression or unacceptable toxicity.

MAINTENANCE: Beginning cycle 5, patients with no evidence of disease after induction receive pembrolizumab IV over 25-40 minutes and gemcitabine intravesically on day 1 of each cycle. Treatment repeats every 3 weeks for 12 cycles in the absence of disease progression or unacceptable toxicity.

Additionally, patients with T1 tumors undergo a re-staging transurethral resection of bladder tumor (TURBT) within 60 days of registration. Patients also undergo urine and blood sample collection, bladder biopsy, cystoscopy, computed tomography (CT) and magnetic resonance imaging (MRI) throughout the study.

After completion of study treatment, patients with evidence of disease (recurrence or progression) or stop study treatment to receive non-protocol treatment during induction are followed up every 6 months for 5 years. Patients who go off treatment due to any reason other than recurrence/progression or receiving subsequent non-protocol treatment during induction will go to clinical follow-up until evidence of disease progression/recurrence. Thereafter, patients are followed up every 6 months until 5 years from registration. Patients who complete scheduled maintenance treatment according to protocol therapy are followed up every 3 months for 2 years and then every 6 months for 3 years until disease progression/recurrence or receiving subsequent non-protocol treatment. Thereafter, patients are followed up every 6 months until 5 years from registration. Patients who have evidence of disease during maintenance therapy are followed up every 6 months until 5 years from registration.

ELIGIBILITY:
Inclusion Criteria:

* High grade Ta, T1 or CIS urothelial carcinoma. Accrual of patients with Ta or T1 disease may be closed to ensure adequate patients enrollment to meet the primary endpoint
* Persistent disease (defined as not achieving disease free status) after completing therapy with at least induction BCG (>= 5 doses) and the first round of maintenance or second induction course (>= 2 doses). The subsequent round of BCG, either maintenance or repeat induction, must be given within 6 months of initial induction BCG
* Persistent high risk NMIBC (T1, high grade Ta and/or CIS) must be within 9 months of the last BCG instillation despite having received adequate BCG as defined above.

  * Registration must be within 12 months of last BCG instillation
* High grade T1 after completing therapy with at least induction BCG (>= 5 doses) or after completing therapy with at least induction BCG (>= 5 doses) and first round of maintenance or second induction course (>= 2 doses). The subsequent round of BCG, either maintenance or repeat induction, must be given within 6 months of initial induction BCG

  * Disease recurrence (T1) must be within 9 months of the last BCG instillation despite having received adequate BCG as defined above
  * Registration must be within 12 months of last BCG instillation
* Mixed variant histology (adenocarcinoma, squamous cell carcinoma) is eligible, but pure variant histology is ineligible
* Patients who are disease free at 6 months after starting BCG but have high grade recurrence (T1, Ta, CIS) while on maintenance therapy would be eligible

  * The recurrence must be within 6 months of the last BCG dose.
  * Registration must be within 12 months of last maintenance BCG instillation
* Patients must be deemed unfit for radical cystectomy by the treating physician or refuse radical cystectomy
* All patients must have histologically confirmed urothelial cancer of the bladder within 60 days prior to registration
* All visible tumor must be completely resected 60 days prior to registration (residual pure CIS is permitted)

  * All patients must have had a cystoscopy (or TURBT with complete resection) without papillary tumor and negative urinary cytology within 28 days of registration (positive cytology is allowed in patients with CIS)
* All patients with T1 tumors must undergo a re-staging transurethral resection of bladder tumor (TURBT) within 60 days of registration

  * There must be uninvolved muscularis propria present in the re-staging TURBT. The initial TURBT prior to re-staging TURBT may be greater than 60 days prior to registration
* Patients must have had imaging with CT or MRI abdomen/pelvis within 90 days of registration demonstrating no evidence of metastasis
* Patients cannot have had a history of urothelial carcinoma in the ureters or prostatic urethra 24 months prior to registration
* Patients must not be currently participating in or have participated in a study of an investigational agent or have used an investigational device within 4 weeks prior to study registration

  * Note: Participants who have entered the follow-up phase of an investigational study may participate as long as it has been more than 4 weeks after the last dose of the previous investigational agent at time of registration
* Patients must not have prior therapy with an anti-PD-1, anti-PD-L1, or anti PD L2 agent or with an agent directed to another stimulatory or co-inhibitory T-cell receptor (e.g., CTLA-4, OX 40, CD137)
* Patients must not have undergone prior allogeneic hematopoietic stem cell transplantation within the last 5 years prior to registration. (Participants who have had a transplant greater than 5 years ago are eligible as long as there are no symptoms of graft versus host disease [GVHD])
* Patients must not have received prior systemic anti-cancer therapy including investigational agents within 4 weeks prior to treatment

  * Note: Participants must have recovered from all adverse events (AEs) due to previous therapies to =< grade 1 or baseline. Participants with =< grade 2 neuropathy may be eligible
  * Note: If participant received major surgery, they must have recovered adequately from the toxicity and/or complications from the intervention prior to starting study treatment
* Patients must not have received prior radiotherapy within 2 weeks of study registration. Participants must have recovered from all radiation-related toxicities, not require corticosteroids, and not have had radiation pneumonitis
* Patients must not have received radiation therapy to the lung that is > 30 Gy within 6 months prior to trial registration
* Not pregnant and not nursing, because this study involves an agent that has known genotoxic, mutagenic and teratogenic effects

  * Women and men of reproductive potential should agree to use an appropriate method of birth control throughout their participation in this study due to the teratogenic potential of the therapy utilized in this trial. Include as applicable: Appropriate methods of birth control include abstinence, oral contraceptives, implantable hormonal contraceptives or double barrier method (diaphragm plus condom)
  * A woman of childbearing potential (WOCBP) must not have a positive urine pregnancy test within 7 days prior to registration. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required
  * Patients must not be pregnant or breastfeeding or expecting to conceive or father children within the projected duration of the study, starting with registration through the last dose of treatment
* Age >= 18 years
* Eastern Cooperative Oncology Group (ECOG) performance status 0-2
* Absolute neutrophil count (ANC) >= 1,500/mm^3
* Platelet count >= 100,000/mm^3
* Hemoglobin >= 9.0 g/dL
* Creatinine =< 1.5 x upper limit of normal (ULN)

  * In patients with creatinine > 1.5 x ULN, if measured or calculated creatinine clearance > 30 mL/min, then patient is eligible
* Total bilirubin =< 1.5 x ULN

  * In patients with a total bilirubin > 1.5 x ULN, if direct bilirubin < 1.0 X ULN, then patient is eligible
* Aspartate aminotransferase (AST)/ alanine aminotransferase (ALT) =< 2.5 x ULN
* Patients must not have had an active autoimmune disease requiring systemic treatment within 24 months prior to registration. Autoimmune diseases include, but not limited to, lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, antiphospholipid syndrome, Wegener's granulomatosis, Sjogren's syndrome, Bell's palsy, Guillain-Barre syndrome, multiple sclerosis, autoimmune thyroid disease, vasculitis, or glomerulonephritis
* Patients must not have a diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy (in dosing exceeding 10 mg daily of prednisone equivalent) or any other form of immunosuppressive therapy within 7 days prior to registration

  * Note: Replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency) is not considered a form of systemic treatment and is allowed
* Patients must not have a known psychiatric or substance abuse disorder that would interfere with the participant's ability to cooperate with the requirements of the study
* Patients must not have active tuberculosis
* Patients must not have been treated with antibiotics for an active infection within 14 days prior to registration. Prophylactic antibiotics are permitted. Treatment for a urinary tract infection (UTI) is allowed but must be deemed adequately treated by the treating physician prior the start of cycle 1 (C1) day 1 (D1)
* Patients must not have a history of idiopathic pulmonary fibrosis or organizing pneumonia
* Patients must not have a history of (non-infectious) pneumonitis that required steroids or have current pneumonitis
* Patients with human immunodeficiency virus (HIV) are eligible with the following:

  * On effective anti-retroviral therapy with undetectable viral load within 6 months of registration
* HIV-infected participants must not have a history of Kaposi sarcoma and/or multicentric Castleman disease
* Patients must not have a known additional malignancy that has had progression or has required active treatment in the last three years. Exceptions include basal or squamous cell carcinoma of the skin that has undergone potentially curative therapy or in situ cervical cancer. A history of prostate cancer that was treated with definitive intent is allowed, provided that the prostate-specific antigen (PSA) is undetectable for at least 1 year while off androgen deprivation therapy
* Patients must not have known active CNS metastases and/or carcinomatous meningitis. Participants with previously treated brain metastases may participate provided they are radiologically stable, i.e., without evidence of progression for at least 4 weeks by repeat imaging (note that the repeat imaging should be performed during study screening), clinically stable and without requirement of steroid treatment for at least 14 days prior to first dose of study treatment
* Patients must not have severe hypersensitivity (>= grade 3) to pembrolizumab and/or any of its excipients
* Patients must not have an active infection requiring systemic therapy
* Patients must not have a known history of hepatitis B (defined as hepatitis B surface antigen [HBsAg] reactive) or known active hepatitis C virus (defined as hepatitis C virus [HCV] ribonucleic acid [RNA] [qualitative] is detected) infection

  * Note: No testing for hepatitis B and hepatitis C is required unless mandated by a local health authority
* Patients must not have received live vaccines within 30 days of study drug administration. Examples of live vaccines include, but are not limited to, the following: measles, mumps, rubella, varicella/zoster (chicken pox), yellow fever, rabies, Bacillus Calmette-Guerin (BCG), and typhoid vaccine. Seasonal influenza vaccines for injection are generally killed virus vaccines and are allowed; however, intranasal influenza vaccines (e.g., FluMist®) are live attenuated vaccines and are not allowed. COVID-19 vaccinations are permitted

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 161 (Estimated)
Dates: Start 2020-03-18 (Actual); Primary Completion 2026-12-09 (Estimated); Study Completion 2026-12-09 (Estimated)

PRIMARY OUTCOMES:
Complete response rate in the carcinoma in situ (CIS) subpopulation | At 6 months (end of cycle 8, week 25)
  A complete response, only for patients with a CIS component, is a cystoscopy without evidence of bladder tumor and negative biopsy (including directed biopsies to any suspicious areas and in addition random bladder biopsies including trigone, left lateral wall, right lateral wall, posterior bladder, dome of bladder, and the prostatic urethra in men), and negative cytology for high grade disease.
Event-free survival at 18 months | From the date of study registration to the first documentation of an event or death whichever comes first, assessed up to 18 months
  For patients without a documented event and who are still alive, they will be censored at last disease assessment. For patients who start any subsequent ant-cancer therapy without any reported events will be censored at their last disease assessment. will be obtained with a Kaplan-Meier estimator (using the Greenwood formula to estimate the variance) for the entire 153 patient group consisting of patients with CIS, CIS with Ta/T1 or Ta or T1 disease. A 90% confidence interval will be generated for the 18-month EFS estimate.

SECONDARY OUTCOMES:
Incidence of adverse events | Up to 5 years post treatment
  Adverse events will be assessed based on the National Cancer Institute common toxicity criteria (Common Terminology Criteria for Adverse Events version 5.0).
Duration of response (DOR) | From the time a patient had a documented response (the time would start at the time a response was first noted) until disease-progression, assessed up to 5 years
  Analysis will only include those patients in the CIS population who achieve a response. Patients who are alive and without a documented progression at the time of analysis will be censored at the time of the last disease status evaluation. The Kaplan-Meier product-limit estimator will be used to estimate DOR, medians and 95% confidence intervals (CI).
Progression-free survival (PFS) | From the date of study registration to the date of progression or death due to any cause, whichever occurs first, assessed up to 5 years
  Surviving patients without any documented progressions will be censored at the date of last known contact. Progression will be defined as the development of muscle invasive bladder cancer or metastatic urothelial cancer (nodal and/or distant). The Kaplan-Meier product-limit estimator will be used to estimate PFS, medians and 95% CI.
Overall survival (OS) | From the date of study registration to date of death due to any cause, assessed up to 5 years
  Surviving patients will be censored at the date of last known contact. The Kaplan-Meier product-limit estimator will be used to estimate OS, medians and 95% CI.
Cystectomy-free survival | From the date of study registration to the date of cystectomy for all patients
  The Kaplan-Meier product-limit estimator will be used to estimate cystectomy-free survival, medians and 95% CI.
Recurrence free survival (RFS) | From the date of study registration to the first documentation of recurrence or death due to any cause, assessed up to 5 years
  Surviving patients without any documented recurrence will be censored at the date of last known contact. Recurrence will be defined as the development of high-grade bladder cancer for patients with a CIS component only and those without a CIS component. The Kaplan-Meier product-limit estimator will be used to estimate RFS, medians and 95% CI.

CONTACTS AND LOCATIONS:
Overall Officials: Michael E Woods, Principal Investigator — Alliance for Clinical Trials in Oncology
Locations (391):
- United States (382):
  - University of Alabama at Birmingham Cancer Center, Birmingham, Alabama
  - Anchorage Associates in Radiation Medicine, Anchorage, Alaska
  - Anchorage Radiation Therapy Center, Anchorage, Alaska
  - Alaska Breast Care and Surgery LLC, Anchorage, Alaska
  - Alaska Oncology and Hematology LLC, Anchorage, Alaska
  - Alaska Women's Cancer Care, Anchorage, Alaska
  - Anchorage Oncology Centre, Anchorage, Alaska
  - Katmai Oncology Group, Anchorage, Alaska
  - Providence Alaska Medical Center, Anchorage, Alaska
  - Fairbanks Memorial Hospital, Fairbanks, Alaska
  - Cancer Center at Saint Joseph's, Phoenix, Arizona
  - Mayo Clinic Hospital in Arizona, Phoenix, Arizona
  - Mayo Clinic in Arizona, Scottsdale, Arizona
  - Mercy Hospital Fort Smith, Fort Smith, Arkansas
  - Providence Saint Joseph Medical Center/Disney Family Cancer Center, Burbank, California
  - Cedars Sinai Medical Center, Los Angeles, California
  - University of California Davis Comprehensive Cancer Center, Sacramento, California
  - Rocky Mountain Cancer Centers-Aurora, Aurora, Colorado
  - The Medical Center of Aurora, Aurora, Colorado
  - Boulder Community Foothills Hospital, Boulder, Colorado
  - Rocky Mountain Cancer Centers-Boulder, Boulder, Colorado
  - Rocky Mountain Cancer Centers - Centennial, Centennial, Colorado
  - Cancer Center of Colorado at Sloan's Lake, Denver, Colorado
  - National Jewish Health-Main Campus, Denver, Colorado
  - The Women's Imaging Center, Denver, Colorado
  - Colorado Blood Cancer Institute, Denver, Colorado
  - Presbyterian - Saint Lukes Medical Center - Health One, Denver, Colorado
  - Rocky Mountain Cancer Centers-Midtown, Denver, Colorado
  - Saint Joseph Hospital - Cancer Centers of Colorado, Denver, Colorado
  - Rocky Mountain Cancer Centers-Rose, Denver, Colorado
  - Rose Medical Center, Denver, Colorado
  - Western Surgical Care, Denver, Colorado
  - Mountain Blue Cancer Care Center - Swedish, Englewood, Colorado
  - Rocky Mountain Cancer Centers - Swedish, Englewood, Colorado
  - Swedish Medical Center, Englewood, Colorado
  - The Melanoma and Skin Cancer Institute, Englewood, Colorado
  - National Jewish Health-Western Hematology Oncology, Golden, Colorado
  - Saint Mary's Hospital and Regional Medical Center, Grand Junction, Colorado
  - Banner North Colorado Medical Center, Greeley, Colorado
  - Good Samaritan Hospital - Cancer Centers of Colorado, Lafayette, Colorado
  - Rocky Mountain Cancer Centers-Lakewood, Lakewood, Colorado
  - Rocky Mountain Cancer Centers-Littleton, Littleton, Colorado
  - Rocky Mountain Cancer Centers-Sky Ridge, Lone Tree, Colorado
  - Sky Ridge Medical Center, Lone Tree, Colorado
  - Banner North Colorado Medical Center - Loveland Campus, Loveland, Colorado
  - National Jewish Health-Northern Hematology Oncology, Thornton, Colorado
  - Rocky Mountain Cancer Centers-Thornton, Thornton, Colorado
  - Intermountain Health Lutheran Hospital, Wheat Ridge, Colorado
  - MedStar Georgetown University Hospital, Washington D.C., District of Columbia
  - MedStar Washington Hospital Center, Washington D.C., District of Columbia
  - Holy Cross Hospital, Fort Lauderdale, Florida
  - UF Health Cancer Institute - Gainesville, Gainesville, Florida
  - Hawaii Cancer Care Inc - Waterfront Plaza, Honolulu, Hawaii
  - Island Urology, Honolulu, Hawaii
  - Queen's Cancer Cenrer - POB I, Honolulu, Hawaii
  - Queen's Medical Center, Honolulu, Hawaii
  - Straub Clinic and Hospital, Honolulu, Hawaii
  - University of Hawaii Cancer Center, Honolulu, Hawaii
  - Hawaii Cancer Care Inc-Liliha, Honolulu, Hawaii
  - Hawaii Diagnostic Radiology Services LLC, Honolulu, Hawaii
  - Kuakini Medical Center, Honolulu, Hawaii
  - Queen's Cancer Center - Kuakini, Honolulu, Hawaii
  - The Cancer Center of Hawaii-Liliha, Honolulu, Hawaii
  - Kapiolani Medical Center for Women and Children, Honolulu, Hawaii
  - Straub Medical Center - Kahului Clinic, Kahului, Hawaii
  - Castle Medical Center, Kailua, Hawaii
  - Wilcox Memorial Hospital and Kauai Medical Clinic, Lihue, Hawaii
  - Hawaii Cancer Care - Westridge, ‘Aiea, Hawaii
  - Pali Momi Medical Center, ‘Aiea, Hawaii
  - Queen's Cancer Center - Pearlridge, ‘Aiea, Hawaii
  - The Cancer Center of Hawaii-Pali Momi, ‘Aiea, Hawaii
  - The Queen's Medical Center - West Oahu, ‘Ewa Beach, Hawaii
  - Saint Alphonsus Cancer Care Center-Boise, Boise, Idaho
  - Saint Luke's Cancer Institute - Boise, Boise, Idaho
  - Saint Alphonsus Cancer Care Center-Caldwell, Caldwell, Idaho
  - Kootenai Health - Coeur d'Alene, Coeur d'Alene, Idaho
  - Walter Knox Memorial Hospital, Emmett, Idaho
  - Saint Luke's Cancer Institute - Fruitland, Fruitland, Idaho
  - Idaho Urologic Institute-Meridian, Meridian, Idaho
  - Saint Luke's Cancer Institute - Meridian, Meridian, Idaho
  - Saint Alphonsus Cancer Care Center-Nampa, Nampa, Idaho
  - Saint Luke's Cancer Institute - Nampa, Nampa, Idaho
  - Kootenai Clinic Cancer Services - Post Falls, Post Falls, Idaho
  - Kootenai Clinic Cancer Services - Sandpoint, Sandpoint, Idaho
  - Saint Luke's Cancer Institute - Twin Falls, Twin Falls, Idaho
  - OSF Saint Anthony's Health Center, Alton, Illinois
  - Illinois CancerCare-Bloomington, Bloomington, Illinois
  - Illinois CancerCare-Canton, Canton, Illinois
  - Memorial Hospital of Carbondale, Carbondale, Illinois
  - SIH Cancer Institute, Carterville, Illinois
  - Illinois CancerCare-Carthage, Carthage, Illinois
  - Centralia Oncology Clinic, Centralia, Illinois
  - Rush MD Anderson Cancer Center, Chicago, Illinois
  - Cancer Care Specialists of Illinois - Decatur, Decatur, Illinois
  - Decatur Memorial Hospital, Decatur, Illinois
  - Illinois CancerCare-Dixon, Dixon, Illinois
  - Crossroads Cancer Center, Effingham, Illinois
  - Illinois CancerCare-Eureka, Eureka, Illinois
  - Illinois CancerCare-Galesburg, Galesburg, Illinois
  - Western Illinois Cancer Treatment Center, Galesburg, Illinois
  - Illinois CancerCare-Kewanee Clinic, Kewanee, Illinois
  - Illinois CancerCare-Macomb, Macomb, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - Marjorie Weinberg Cancer Center at Loyola-Gottlieb, Melrose Park, Illinois
  - SSM Health Good Samaritan, Mount Vernon, Illinois
  - Cancer Care Center of O'Fallon, O'Fallon, Illinois
  - Illinois CancerCare-Ottawa Clinic, Ottawa, Illinois
  - Illinois CancerCare-Pekin, Pekin, Illinois
  - Illinois CancerCare-Peoria, Peoria, Illinois
  - Methodist Medical Center of Illinois, Peoria, Illinois
  - Illinois CancerCare-Peru, Peru, Illinois
  - Valley Radiation Oncology, Peru, Illinois
  - Illinois CancerCare-Princeton, Princeton, Illinois
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - Springfield Clinic, Springfield, Illinois
  - Springfield Memorial Hospital, Springfield, Illinois
  - Southwest Illinois Health Services LLP, Swansea, Illinois
  - Illinois CancerCare - Washington, Washington, Illinois
  - Reid Health, Richmond, Indiana
  - Memorial Hospital of South Bend, South Bend, Indiana
  - Central Care Cancer Center - Garden City, Garden City, Kansas
  - Central Care Cancer Center - Great Bend, Great Bend, Kansas
  - University of Kansas Cancer Center, Kansas City, Kansas
  - University of Kansas Hospital-Indian Creek Campus, Overland Park, Kansas
  - University of Kansas Hospital-Westwood Cancer Center, Westwood, Kansas
  - University of Kentucky/Markey Cancer Center, Lexington, Kentucky
  - Louisiana Hematology Oncology Associates LLC, Baton Rouge, Louisiana
  - Mary Bird Perkins Cancer Center, Baton Rouge, Louisiana
  - Mary Bird Perkins Cancer Center - Metairie, Metairie, Louisiana
  - East Jefferson General Hospital, Metairie, Louisiana
  - LSU Healthcare Network / Metairie Multi-Specialty Clinic, Metairie, Louisiana
  - Louisiana State University Health Science Center, New Orleans, Louisiana
  - University Medical Center New Orleans, New Orleans, Louisiana
  - Touro Infirmary, New Orleans, Louisiana
  - UM Baltimore Washington Medical Center/Tate Cancer Center, Glen Burnie, Maryland
  - Lowell General Hospital, Lowell, Massachusetts
  - Mercy Medical Center, Springfield, Massachusetts
  - Hickman Cancer Center, Adrian, Michigan
  - Trinity Health Saint Joseph Mercy Hospital Ann Arbor, Ann Arbor, Michigan
  - Bronson Battle Creek, Battle Creek, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology - Brighton, Brighton, Michigan
  - Trinity Health Medical Center - Brighton, Brighton, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology - Canton, Canton, Michigan
  - Trinity Health Medical Center - Canton, Canton, Michigan
  - Caro Cancer Center, Caro, Michigan
  - Chelsea Hospital, Chelsea, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology - Chelsea Hospital, Chelsea, Michigan
  - Hematology Oncology Consultants-Clarkston, Clarkston, Michigan
  - Newland Medical Associates-Clarkston, Clarkston, Michigan
  - Henry Ford Health Saint John Hospital, Detroit, Michigan
  - Henry Ford River District Hospital, East China Township, Michigan
  - Cancer Hematology Centers - Flint, Flint, Michigan
  - Genesee Hematology Oncology PC, Flint, Michigan
  - Genesys Hurley Cancer Institute, Flint, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Corewell Health Grand Rapids Hospitals - Butterworth Hospital, Grand Rapids, Michigan
  - Corewell Health Grand Rapids Hospitals - Helen DeVos Children's Hospital, Grand Rapids, Michigan
  - Trinity Health Grand Rapids Hospital, Grand Rapids, Michigan
  - Henry Ford Saint John Hospital - Academic, Grosse Pointe Woods, Michigan
  - Henry Ford Saint John Hospital - Breast, Grosse Pointe Woods, Michigan
  - Henry Ford Saint John Hospital - Van Elslander, Grosse Pointe Woods, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Beacon Kalamazoo Cancer Center, Kalamazoo, Michigan
  - Beacon Kalamazoo, Kalamazoo, Michigan
  - University of Michigan Health - Sparrow Lansing, Lansing, Michigan
  - Hope Cancer Clinic, Livonia, Michigan
  - Trinity Health Saint Mary Mercy Livonia Hospital, Livonia, Michigan
  - Henry Ford Saint John Hospital - Macomb Medical, Macomb, Michigan
  - Henry Ford Warren Hospital - Breast Macomb, Macomb, Michigan
  - Saint Mary's Oncology/Hematology Associates of Marlette, Marlette, Michigan
  - Toledo Clinic Cancer Centers-Monroe, Monroe, Michigan
  - Trinity Health Muskegon Hospital, Muskegon, Michigan
  - Corewell Health Lakeland Hospitals - Niles Hospital, Niles, Michigan
  - Cancer and Hematology Centers of Western Michigan - Norton Shores, Norton Shores, Michigan
  - Hope Cancer Center, Pontiac, Michigan
  - Michigan Healthcare Professionals Pontiac, Pontiac, Michigan
  - Newland Medical Associates-Pontiac, Pontiac, Michigan
  - Trinity Health Saint Joseph Mercy Oakland Hospital, Pontiac, Michigan
  - Corewell Health Reed City Hospital, Reed City, Michigan
  - Henry Ford Rochester Hospital, Rochester Hills, Michigan
  - MyMichigan Medical Center Saginaw, Saginaw, Michigan
  - Oncology Hematology Associates of Saginaw Valley PC, Saginaw, Michigan
  - Corewell Health Lakeland Hospitals - Marie Yeager Cancer Center, Saint Joseph, Michigan
  - Corewell Health Lakeland Hospitals - Saint Joseph Hospital, Saint Joseph, Michigan
  - Bhadresh Nayak MD PC-Sterling Heights, Sterling Heights, Michigan
  - MyMichigan Medical Center Tawas, Tawas City, Michigan
  - Munson Medical Center, Traverse City, Michigan
  - Advanced Breast Care Center PLLC, Warren, Michigan
  - Henry Ford Health Warren Hospital, Warren, Michigan
  - Henry Ford Madison Heights Hospital - Breast, Warren, Michigan
  - Henry Ford Warren Hospital - GLCMS, Warren, Michigan
  - Macomb Hematology Oncology PC, Warren, Michigan
  - Saint Mary's Oncology/Hematology Associates of West Branch, West Branch, Michigan
  - University of Michigan Health - West, Wyoming, Michigan
  - Huron Gastroenterology PC, Ypsilanti, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology Ann Arbor Campus, Ypsilanti, Michigan
  - Fairview Ridges Hospital, Burnsville, Minnesota
  - Minnesota Oncology - Burnsville, Burnsville, Minnesota
  - Cambridge Medical Center, Cambridge, Minnesota
  - Mercy Hospital, Coon Rapids, Minnesota
  - Fairview Southdale Hospital, Edina, Minnesota
  - Unity Hospital, Fridley, Minnesota
  - Fairview Clinics and Surgery Center Maple Grove, Maple Grove, Minnesota
  - Minnesota Oncology Hematology PA-Maplewood, Maplewood, Minnesota
  - Saint John's Hospital - Healtheast, Maplewood, Minnesota
  - Abbott-Northwestern Hospital, Minneapolis, Minnesota
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - Health Partners Inc, Minneapolis, Minnesota
  - Monticello Cancer Center, Monticello, Minnesota
  - New Ulm Medical Center, New Ulm, Minnesota
  - Fairview Northland Medical Center, Princeton, Minnesota
  - North Memorial Medical Health Center, Robbinsdale, Minnesota
  - Park Nicollet Clinic - Saint Louis Park, Saint Louis Park, Minnesota
  - Regions Hospital, Saint Paul, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - Saint Francis Regional Medical Center, Shakopee, Minnesota
  - Lakeview Hospital, Stillwater, Minnesota
  - Ridgeview Medical Center, Waconia, Minnesota
  - Rice Memorial Hospital, Willmar, Minnesota
  - Minnesota Oncology Hematology PA-Woodbury, Woodbury, Minnesota
  - Fairview Lakes Medical Center, Wyoming, Minnesota
  - Mercy Oncology and Hematology - Clayton-Clarkson, Ballwin, Missouri
  - Central Care Cancer Center - Bolivar, Bolivar, Missouri
  - Cox Cancer Center Branson, Branson, Missouri
  - Mercy Cancer Center - Cape Girardeau, Cape Girardeau, Missouri
  - Saint Francis Medical Center, Cape Girardeau, Missouri
  - Saint Luke's Hospital, Chesterfield, Missouri
  - MU Health - University Hospital/Ellis Fischel Cancer Center, Columbia, Missouri
  - Parkland Health Center - Farmington, Farmington, Missouri
  - MU Health Care Goldschmidt Cancer Center, Jefferson City, Missouri
  - Freeman Health System, Joplin, Missouri
  - Mercy Hospital Joplin, Joplin, Missouri
  - Mercy Clinic-Rolla-Cancer and Hematology, Rolla, Missouri
  - Phelps Health Delbert Day Cancer Institute, Rolla, Missouri
  - Heartland Regional Medical Center, Saint Joseph, Missouri
  - Sainte Genevieve County Memorial Hospital, Sainte Genevieve, Missouri
  - Mercy Hospital Springfield, Springfield, Missouri
  - CoxHealth South Hospital, Springfield, Missouri
  - Mercy Infusion Center - Chippewa, St Louis, Missouri
  - Mercy Hospital South, St Louis, Missouri
  - Missouri Baptist Medical Center, St Louis, Missouri
  - Mercy Hospital Saint Louis, St Louis, Missouri
  - Missouri Baptist Sullivan Hospital, Sullivan, Missouri
  - BJC Outpatient Center at Sunset Hills, Sunset Hills, Missouri
  - Mercy Hospital Washington, Washington, Missouri
  - Community Hospital of Anaconda, Anaconda, Montana
  - Billings Clinic Cancer Center, Billings, Montana
  - Saint Vincent Healthcare, Billings, Montana
  - Saint Vincent Frontier Cancer Center, Billings, Montana
  - Bozeman Health Deaconess Hospital, Bozeman, Montana
  - Saint James Community Hospital and Cancer Treatment Center, Butte, Montana
  - Benefis Sletten Cancer Institute, Great Falls, Montana
  - Great Falls Clinic, Great Falls, Montana
  - Logan Health Medical Center, Kalispell, Montana
  - Saint Patrick Hospital - Community Hospital, Missoula, Montana
  - Community Medical Center, Missoula, Montana
  - Dartmouth Hitchcock Medical Center/Dartmouth Cancer Center, Lebanon, New Hampshire
  - Memorial Sloan Kettering Basking Ridge, Basking Ridge, New Jersey
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Memorial Sloan Kettering Monmouth, Middletown, New Jersey
  - Memorial Sloan Kettering Bergen, Montvale, New Jersey
  - The Valley Hospital - Luckow Pavilion, Paramus, New Jersey
  - Neurosurgeons of New Jersey-Ridgewood, Ridgewood, New Jersey
  - Valley Health System Ridgewood Campus, Ridgewood, New Jersey
  - Valley Health System-Hematology/Oncology, Westwood, New Jersey
  - Memorial Sloan Kettering Commack, Commack, New York
  - Arnot Ogden Medical Center/Falck Cancer Center, Elmira, New York
  - The New York Hospital Medical Center of Queens, Flushing, New York
  - Memorial Sloan Kettering Westchester, Harrison, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - NYP/Weill Cornell Medical Center, New York, New York
  - Stony Brook University Medical Center, Stony Brook, New York
  - Memorial Sloan Kettering Nassau, Uniondale, New York
  - UNC Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina
  - University of North Carolina-Hillsborough Campus, Hillsborough, North Carolina
  - Indu and Raj Soin Medical Center, Beavercreek, Ohio
  - Saint Elizabeth Boardman Hospital, Boardman, Ohio
  - Dayton Physicians LLC-Miami Valley South, Centerville, Ohio
  - Miami Valley Hospital South, Centerville, Ohio
  - Oncology Hematology Care Inc-Kenwood, Cincinnati, Ohio
  - Miami Valley Hospital, Dayton, Ohio
  - Dayton Physician LLC - Englewood, Dayton, Ohio
  - Miami Valley Hospital North, Dayton, Ohio
  - Armes Family Cancer Center, Findlay, Ohio
  - Blanchard Valley Hospital, Findlay, Ohio
  - Orion Cancer Care, Findlay, Ohio
  - Atrium Medical Center-Middletown Regional Hospital, Franklin, Ohio
  - Dayton Physicians LLC-Atrium, Franklin, Ohio
  - Dayton Physicians LLC-Wayne, Greenville, Ohio
  - Wayne Hospital, Greenville, Ohio
  - Greater Dayton Cancer Center, Kettering, Ohio
  - First Dayton Cancer Care, Kettering, Ohio
  - Kettering Medical Center, Kettering, Ohio
  - Mercy Health - Perrysburg Hospital, Perrysburg, Ohio
  - Springfield Regional Cancer Center, Springfield, Ohio
  - Springfield Regional Medical Center, Springfield, Ohio
  - Mercy Health - Saint Anne Hospital, Toledo, Ohio
  - Toledo Clinic Cancer Centers-Toledo, Toledo, Ohio
  - Dayton Physicians LLC - Troy, Troy, Ohio
  - Upper Valley Medical Center, Troy, Ohio
  - Saint Joseph Warren Hospital, Warren, Ohio
  - Saint Elizabeth Youngstown Hospital, Youngstown, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Mercy Hospital Oklahoma City, Oklahoma City, Oklahoma
  - Saint Alphonsus Cancer Care Center-Baker City, Baker City, Oregon
  - Saint Charles Health System, Bend, Oregon
  - Clackamas Radiation Oncology Center, Clackamas, Oregon
  - Providence Cancer Institute Clackamas Clinic, Clackamas, Oregon
  - Bay Area Hospital, Coos Bay, Oregon
  - Providence Newberg Medical Center, Newberg, Oregon
  - Saint Alphonsus Cancer Care Center-Ontario, Ontario, Oregon
  - Providence Portland Medical Center, Portland, Oregon
  - Providence Saint Vincent Medical Center, Portland, Oregon
  - Saint Charles Health System-Redmond, Redmond, Oregon
  - Lehigh Valley Hospital-Cedar Crest, Allentown, Pennsylvania
  - Lehigh Valley Hospital - Muhlenberg, Bethlehem, Pennsylvania
  - Pocono Medical Center, East Stroudsburg, Pennsylvania
  - Lehigh Valley Hospital-Hazleton, Hazleton, Pennsylvania
  - Ralph H Johnson VA Medical Center, Charleston, South Carolina
  - Gibbs Cancer Center-Gaffney, Gaffney, South Carolina
  - Gibbs Cancer Center-Pelham, Greer, South Carolina
  - North Grove Medical Park, Spartanburg, South Carolina
  - Spartanburg Medical Center, Spartanburg, South Carolina
  - Spartanburg Medical Center - Mary Black Campus, Spartanburg, South Carolina
  - SMC Center for Hematology Oncology Union, Union, South Carolina
  - University of Texas Medical Branch, Galveston, Texas
  - Baylor College of Medicine/Dan L Duncan Comprehensive Cancer Center, Houston, Texas
  - UTMB Cancer Center at Victory Lakes, League City, Texas
  - Audie L Murphy VA Hospital, San Antonio, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - American Fork Hospital / Huntsman Intermountain Cancer Center, American Fork, Utah
  - Sandra L Maxwell Cancer Center, Cedar City, Utah
  - Logan Regional Hospital, Logan, Utah
  - Intermountain Medical Center, Murray, Utah
  - McKay-Dee Hospital Center, Ogden, Utah
  - Utah Valley Regional Medical Center, Provo, Utah
  - Riverton Hospital, Riverton, Utah
  - Utah Cancer Specialists-Salt Lake City, Salt Lake City, Utah
  - LDS Hospital, Salt Lake City, Utah
  - Saint George Regional Medical Center, St. George, Utah
  - Providence Regional Cancer System-Aberdeen, Aberdeen, Washington
  - MultiCare Auburn Medical Center, Auburn, Washington
  - PeaceHealth Saint Joseph Medical Center, Bellingham, Washington
  - Providence Regional Cancer System-Centralia, Centralia, Washington
  - Swedish Cancer Institute-Edmonds, Edmonds, Washington
  - Providence Regional Cancer Partnership, Everett, Washington
  - MultiCare Gig Harbor Medical Park, Gig Harbor, Washington
  - Swedish Cancer Institute-Issaquah, Issaquah, Washington
  - Kadlec Clinic Hematology and Oncology, Kennewick, Washington
  - Providence Regional Cancer System-Lacey, Lacey, Washington
  - PeaceHealth Saint John Medical Center, Longview, Washington
  - Jefferson Healthcare, Port Townsend, Washington
  - MultiCare Good Samaritan Hospital, Puyallup, Washington
  - Pacific Gynecology Specialists, Seattle, Washington
  - Swedish Medical Center-Ballard Campus, Seattle, Washington
  - Swedish Medical Center-Cherry Hill, Seattle, Washington
  - Swedish Medical Center-First Hill, Seattle, Washington
  - PeaceHealth United General Medical Center, Sedro-Woolley, Washington
  - Providence Regional Cancer System-Shelton, Shelton, Washington
  - MultiCare Deaconess Cancer and Blood Specialty Center - Downtown, Spokane, Washington
  - MultiCare Deaconess Cancer and Blood Specialty Center - North, Spokane, Washington
  - MultiCare Deaconess Cancer and Blood Specialty Center - Valley, Spokane Valley, Washington
  - MultiCare Tacoma General Hospital, Tacoma, Washington
  - PeaceHealth Southwest Medical Center, Vancouver, Washington
  - Providence Saint Mary Regional Cancer Center, Walla Walla, Washington
  - Providence Regional Cancer System-Yelm, Yelm, Washington
  - Marshfield Medical Center-EC Cancer Center, Eau Claire, Wisconsin
  - Marshfield Medical Center-Marshfield, Marshfield, Wisconsin
  - Medical College of Wisconsin, Milwaukee, Wisconsin
  - Marshfield Medical Center - Minocqua, Minocqua, Wisconsin
  - ProHealth D N Greenwald Center, Mukwonago, Wisconsin
  - Cancer Center of Western Wisconsin, New Richmond, Wisconsin
  - ProHealth Oconomowoc Memorial Hospital, Oconomowoc, Wisconsin
  - Marshfield Medical Center-Rice Lake, Rice Lake, Wisconsin
  - Marshfield Medical Center-River Region at Stevens Point, Stevens Point, Wisconsin
  - ProHealth Waukesha Memorial Hospital, Waukesha, Wisconsin
  - UW Cancer Center at ProHealth Care, Waukesha, Wisconsin
  - Marshfield Medical Center - Weston, Weston, Wisconsin
  - Cheyenne Regional Medical Center-West, Cheyenne, Wyoming
  - Billings Clinic-Cody, Cody, Wyoming
  - Welch Cancer Center, Sheridan, Wyoming
- FHP Health Center-Guam, Tamuning, Guam
- Puerto Rico (8):
  - Cancer Center-Metro Medical Center Bayamon, Bayamón
  - Puerto Rico Hematology Oncology Group, Bayamón
  - HIMA San Pablo Oncologic Hospital, Caguas
  - Doctors Cancer Center, Manatí
  - Instituto Oncologia Moderna Ponce, Ponce
  - San Juan Community Oncology Group, San Juan
  - Centro Comprensivo de Cancer de UPR, San Juan
  - San Juan City Hospital, San Juan

IPD SHARING:
Plan to Share IPD: Yes
NCI is committed to sharing data in accordance with NIH policy. For more details on how clinical trial data is shared, access the link to the NIH data sharing policy page.
URL: https://grants.nih.gov/policy/sharing.htm